CLINICAL TRIAL: NCT00233922
Title: Reconstruction of the Orbit With a Bioresorbable Polycaprolactone Implant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National Healthcare Group, Singapore (Other Government)
Responsible Party: Thiam-Chye Lim, MBBS, FRCS, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHG/RPR/04024; NHG/RPR/04024
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Orbital Trauma; Orbital Fractures
Keywords: orbit; orbital; trauma; fractures; facial
MeSH Terms: conditions — Orbital Fractures; Wounds and Injuries; Fractures, Bone; Facies

INTERVENTIONS:
Device: Osteosheet(r)

SUMMARY:
Patients with orbital injuries are entered into the trial. Age: 20 - 70. After obtaining appropriate consent, they are entered into either a control arm where reconstruction of the orbit is done with a titanium mesh (established practice) or the experimental arm where reconstruction is by a bioresorbable implant made of polycaprolactone. Patients are followuped at 1 week, 1 month, 3 months, 6 months & 12 months. CT scan of the orbits are performed preop, 6 months & 12 months. End point is the 12 month follow-up appointment. Visual acuity, range of motion, enophthalmos & diplopia are assessed in follow-up.

DETAILED DESCRIPTION:
Patients with orbital injuries are entered into the trial. Age: 20 - 70. After obtaining appropriate consent, they are entered into either a control arm where reconstruction of the orbit is done with a titanium mesh (established practice) or the experimental arm where reconstruction is by a bioresorbable implant made of polycaprolactone. Patients are followuped at 1 week, 1 month, 3 months, 6 months & 12 months. CT scan of the orbits are performed preop, 6 months & 12 months. End point is the 12 month follow-up appointment. Visual acuity, range of motion, enophthalmos & diplopia are assessed in follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age: 20 - 70 years facial trauma with orbital fractures

Exclusion Criteria:

* No other coexistent conditions eg. diabetes, heart disease, etc

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2004-07; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
visual acuity
Enophthalmos
Diplopia
Cosmetic appearance

CONTACTS AND LOCATIONS:
Overall Officials: Thiam-Chye Lim, MBBS, FRCS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore